CLINICAL TRIAL: NCT05525572
Title: Combining Shockwave Therapy and Platelet Rich Plasma to Treat Erectile Dysfunction in Diabetic Men (COCKTAIL-DM)
Acronym: COCKTAIL-DM
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Funding ended
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Thomas Masterson, Assistant Professor, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20220540
Record Dates: First submitted 2022-04-13; First posted 2022-09-01 (Actual); Results first posted 2025-02-28 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Erectile Dysfunction With Diabetes Mellitus
MeSH Terms: interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Shockwave Therapy (SWT) + Platelet-Rich Plasma (PRP) Group (Experimental): Participants will receive a combination of 5 weekly extracorporeal shockwave therapy sessions (SWT) and two sessions of autologous platelet-rich plasma (PRP) penile injection.
  Interventions: Device: Shockwave Therapy (SWT); Drug: Autologous Platelet-Rich Plasma (PRP)

INTERVENTIONS:
Device: Shockwave Therapy (SWT) — Shockwave Therapy (SWT):
  720 shocks will be administered administered in every session to each treated region (left and right corpora cavernosa and crura). Each session will last approximately 20 minutes. A total of 3600 shocks will be administered over 5 weekly sessions.
Drug: Autologous Platelet-Rich Plasma (PRP) — Autologous Platelet Rich Plasma (PRP):
  5 mL PRP will be administered via intra-cavernous penile injection with a 30 ± 7 day treatment interval.

SUMMARY:
The purpose of this research study is to evaluate whether the combination of Shockwave Therapy (SWT) with Platelet Rich Plasma (PRP) is synergistic and can reverse the pathology of microvascular Erectile Dysfunction (ED) and enhance erectile function in diabetics patients.

ELIGIBILITY:
Inclusion Criteria:

1. Male
2. Between 30 to 80 years of age (inclusive).
3. Be able to provide written informed consent.
4. Have a diagnosis of Mild to Moderate ED (12-21) or Mild ED (22-25) based on International Index of Erectile Dysfunction - Erectile Function (IIEF-EF) questionnaire score.
5. Have diagnosis of Diabetes Mellitus (Type 1 or Type 2), as documented by history of Hemoglobin A1C > 7% OR on medical therapy for Diabetes.
6. Be in a stable relationship and have a minimum of 2 sexual attempts per month for at least one month prior to enrollment.
7. Agree to comply with all study related tests/procedures.

Exclusion Criteria:

1. Previous penile surgery of any kind (except circumcision and condyloma removal), such as penile lengthening, penile cancer surgery, penile plication, grafting.
2. Previous history of priapism, penile fracture, Peyronie's Disease, or penile curvature that negatively influences sexual activity.
3. Abnormal morning serum testosterone level defined as a value lower than 300 ng/dL (±5%).
4. Psychogenic ED as determined by study investigator.
5. Patients using Intracavernous Injections (ICI) for management of ED.
6. Patients with generalized polyneuropathy, neurological conditions, or psychiatric disease (such as bipolar disorder or depression).
7. Have a serious comorbid illness or condition that, in the opinion of the investigator, may compromise the safety or compliance of the subject or preclude successful completion of the study.
8. History of consistent treatment failure with Phosphodiesterase 5 (PDE5) inhibitors for therapy of ED.
9. Poorly controlled diabetes as indicated by Hemoglobin a1c > 7.5%.
10. Use of antiplatelet medications

Ages: 30 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2024-02-12 (Actual); Primary Completion 2024-08-02 (Actual); Study Completion 2024-08-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas A Masterson, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, School of Medicine - Desai Sethi Urology Institute, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Shockwave Therapy (SWT) + Platelet-Rich Plasma (PRP) Group: Participants will receive a combination of 5 weekly extracorporeal shockwave therapy sessions (SWT) and two sessions of autologous platelet-rich plasma (PRP) penile injection.
  Shockwave Therapy (SWT): Shockwave Therapy (SWT):
  720 shocks will be administered administered in every session to each treated region (left and right corpora cavernosa and crura). Each session will last approximately 20 minutes. A total of 3600 shocks will be administered over 5 weekly sessions.
  Autologous Platelet-Rich Plasma (PRP): Autologous Platelet Rich Plasma (PRP):
  5 mL PRP will be administered via intra-cavernous penile injection with a 30 ± 7 day treatment interval.
Period: Overall Study
Arm/Group | Shockwave Therapy (SWT) + Platelet-Rich Plasma (PRP) Group
Started | 2
Completed | 0
Not Completed | 2
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Arm/Group | Shockwave Therapy (SWT) + Platelet-Rich Plasma (PRP) Group
Number analyzed (Participants) | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Markers of Vasodilation
Description: Markers of vasodilation including Endothelial Nitric Oxide Synthase (eNOS) and Neuronal Nitric Oxide Synthase (nNOS) will be measured from serum blood samples in units of ug/mL.
Time Frame: Baseline, Month 3, Month 6
Population: Baseline blood samples unusable due to hemolysis and low cell recovery. Follow up data was not collected due to lost to follow up.
Arm/Group | Shockwave Therapy (SWT) + Platelet-Rich Plasma (PRP) Group
Number analyzed (Participants) | 0

2. Primary Outcome: Endothelial Function Markers
Description: Markers of endothelial function will include Vascular Endothelial Growth Factor (VEGF), Stromal cell-derived factor 1 (SDF-1α), and Stem Cell Factor (SCF). All measured from serum blood samples in units of pg/mL.
Time Frame: Baseline, Month 3, Month 6
Population: as for outcome 1
Arm/Group | Shockwave Therapy (SWT) + Platelet-Rich Plasma (PRP) Group
Number analyzed (Participants) | 0

3. Primary Outcome: Markers of Neo-angiogenesis
Description: Markers of neo-angiogenesis reported as the percentage of Cluster of Differentiation 31 positive cells (CD31+), as measured from serum blood samples and expressed as a percentage.
Time Frame: Baseline to Month 3, Baseline to Month 6
Population: as for outcome 1
Arm/Group | Shockwave Therapy (SWT) + Platelet-Rich Plasma (PRP) Group
Number analyzed (Participants) | 0

4. Primary Outcome: Endothelial Progenitor Cell Colony Forming Units (EPC-CFUs)
Description: Endothelial Progenitor Cell (EPC) Colony Forming Units (CFUs) as measured from peripheral blood samples in units of average cells per well.
Time Frame: Baseline, Month 3, Month 6
Population: Baseline blood samples unusable due to low cell recovery. Follow up data was not collected due to lost to follow up.
Arm/Group | Shockwave Therapy (SWT) + Platelet-Rich Plasma (PRP) Group
Number analyzed (Participants) | 0

5. Secondary Outcome: Penile Blood Flow
Description: Penile Blood Flow will be reported as Peak Systolic Velocity (PSV) and End Diastolic Velocity (EDV), both assessed in cm/sec, via Penile Doppler ultrasonography.
Time Frame: Baseline
Population: First subject completed baseline ultrasound. Second subject did not complete baseline ultrasound. Both subjects were lost to follow up before completing the month 6 visit. The measured value for Right EDV is "0.0", not a missing value.
Measure: Mean (Standard Deviation); unit: cm/sec
Arm/Group | Shockwave Therapy (SWT) + Platelet-Rich Plasma (PRP) Group
Number analyzed (Participants) | 1
cm/sec
  Right Peak Systolic Velocity (PSV) | 39.1
  Right End Diastolic Velocity (EDV) | 0.0
  Left Peak Systolic Velocity (PSV) | 35.4
  Left End Diastolic Velocity (EDV) | 4.2

6. Secondary Outcome: EDITS Questionnaire Scores
Description: Treatment satisfaction is assessed by the Erectile Dysfunction Inventory of Treatment Satisfaction (EDITS) questionnaire. EDITS questionnaire is an 11-item tool addressing participant satisfaction with ED therapy. Each item is a 5-point Likert-type scale from 0 "no satisfaction or dissatisfaction" to 4 "high satisfaction." Total scoring ranges from 0-44 with higher scores indicating higher treatment satisfaction.
Time Frame: Month 3 and Month 6
Population: Data was not collected due to lost to follow up
Arm/Group | Shockwave Therapy (SWT) + Platelet-Rich Plasma (PRP) Group
Number analyzed (Participants) | 0

7. Secondary Outcome: Incidence of Serious Adverse Events (SAEs)
Description: Incidence of Serious Adverse Events (SAEs), as assessed by study physician.
Time Frame: Baseline, up to 6 months
Population: Both subjects were considered "lost to follow up" after completing baseline and Day 0 (treatment visit #1).
Measure: Number; unit: events
Arm/Group | Shockwave Therapy (SWT) + Platelet-Rich Plasma (PRP) Group
Number analyzed (Participants) | 2
events | 0

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Shockwave Therapy (SWT) + Platelet-Rich Plasma (PRP) Group
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-06-27): https://cdn.clinicaltrials.gov/large-docs/72/NCT05525572/Prot_SAP_000.pdf